CLINICAL TRIAL: NCT03363217
Title: A Phase 2 Study of Trametinib for Patients With Pediatric Glioma or Plexiform Neurofibroma With Refractory Tumor and Activation of the MAPK/ERK Pathway.
Brief Title: Trametinib for Pediatric Neuro-oncology Patients With Refractory Tumor and Activation of the MAPK/ERK Pathway.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Montreal Children's Hospital of the MUHC (Other); CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Dr Perreault, Principal Investigator, St. Justine's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Trametinib study TRAM-01
Record Dates: First submitted 2017-11-10; First posted 2017-12-06 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Low-grade Glioma; Plexiform Neurofibroma; Central Nervous System Glioma
Keywords: Glioma; Optic Pathway Glioma; Low grade glioma; MAPK/ERK; Plexiform Neurofibroma; Neurofibromatosis Type 1; Central Nervous System; CNS; Brain Tumor; LGG; NF1; KIAA1549-BRAF; Mitogen-activated Protein Kinase (MEK) inhibitor; Trametinib
MeSH Terms: conditions — Neurofibroma, Plexiform; Glioma; Neurofibromatosis 1; Brain Neoplasms | interventions — trametinib

STUDY DESIGN:
Intervention Model Description: This trial will include 4 parallel groups. Each group will include a particular type of peripheral nerve or central nervous system tumor or mutation.
Masking Description: There is no masking as part of this study. Only one study treatment will be given to all treatment groups at age and weight based dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Neurofibromatosis Type 1 (NF1) with low-grade glioma (Experimental): Patients presenting with Neurofibromatosis Type 1 (NF1) and a progressing/refractory low-grade glioma.
  Interventions: Drug: Trametinib
- Neurofibromatosis Type 1 (NF1) with Plexiform Neurofibroma (Experimental): Patients presenting with Neurofibromatosis Type 1 (NF1) and a plexiform neurofibroma
  Interventions: Drug: Trametinib
- Progressing/refractory low grade-glioma, KIAA1549-BRAF fusion (Experimental): Patients presenting with a progressing/refractory low-grade glioma with a KIAA1549-BRAF fusion.
  Interventions: Drug: Trametinib
- Progressing/Refractory central nervous system (CNS) glioma. (Experimental): Patients presenting with a progressing/refractory central nervous system glioma with an activation of the MAPK/ERK pathway who do not meet criteria for inclusion in other study groups.
  Interventions: Drug: Trametinib

INTERVENTIONS:
Drug: Trametinib — Daily administration of oral trametinib at a unique dose of 0.025 mg/kg.
  Other Names: Mekinist

SUMMARY:
This is a phase 2, open-label, interventional clinical trial that will study the response rate of pediatric glioma and plexiform neurofibroma (PN) to oral administration of trametinib. Patients meeting all inclusion criteria for a given study group will receive the study medication at a daily dose of 0.025 mg/kg up to a total of 18 cycles, in 28-day cycles. A total of 150 patients will be recruited as part of this clinical study.

Patients aged between 1 month (corrected age) and 25 years old will be eligible, in order to include a maximum of patients affected by low-grade glioma (LGG) and PN. This study includes four groups: patients with neurofibromatosis type 1 (NF1) and LGG, NF1 patients with PN, patients with LGG with a B-Raf Serine/Threonine-protein Kinase/Proto-oncogene Encoding B-Raf (BRAF) fusion and patients with glioma of any grade with activation of the Mitogen-activated Protein Kinase/Extracellular Signal-regulated Kinases (MAPK/ERK) pathway. All patients except patients with PN must have failed at least one line of treatment.

The study will also explore the molecular mechanisms behind tumor development, progression and resistance to treatment. Furthermore, this study will also explore important aspects for patients with brain tumors by including assessment of quality of life and neuropsychological evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent Prior to study participation, written informed consent from participants, or in the case of minors, written permission (informed consent) from parents, guardians, or legally acceptable representatives must be obtained according to local laws and regulations.
2. Assent Assent from minor participants should be obtained per local laws and regulations and should be documented in accordance with local requirements.
3. Study activities compliance. Participants must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study, including disease assessment by contrast-enhanced MRI.
4. Age Patient must be aged ≥ 1 month (corrected age) to ≤ 25 years when starting trametinib.
5. Study group Participants must belong to one of the following groups to be eligible. Group 1: NF1 with progressing/refractory LGG Group 2: NF1 with PN Group 3: Progressing/refractory LGG with KIAA 1549-BRAF fursion Group 4: Progressing/refractory glioma with activation of the MPAK/ERK pathway who do not meet criteria for other study groups
6. Tumor Tissue Sample Tumor tissue will be required for all patients (minimally paraffin-embedded tissue block and additionally fresh frozen tissue [if available]). Patients with NF1 and LGG or PN can still be enrolled without tissue if no surgery or biopsy was conducted.

7 Previous MRI At least two previous MRIS fro Group 1, 3, 4 and one previous MRI for Group 2 must be available for central review.

8. Prior therapy Participants must have failed at least one line of treatment including chemotherapy and/or radiation therapy except for plexiform neurofibroma (since there is no recognized standard treatment for his tumor).

9. Prior therapy toxicity Patients must have recovered to grade ≤ 1 from acute toxic effects of all prior chemotherapy, immunotherapy or radiotherapy prior to enrollment except for alopecia and non-treatment related clinically insignificant laboratory abnormalities. prior to starting trametinib. Toxicities will be graded as per the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version 5.0

10. Prior therapy timeline Participants having previously received a chemotherapy agent(s) and/or radiation must conform to the timeline described below. There is no limitation on the number of previous treatments or cycles received.

* An interval of at least 28 days after the last dose of a myelosuppressive chemotherapy, and at least 42 days after the last dose of Nitrosoureas is required prior to starting trametinib.
* An interval of at least 28 days after the last dose of any biologic agents including monoclonal antibody treatment, immunotherapy, viral therapy and other investigational agent is required prior to starting trametinib.
* An interval of at least 84 days after the end of the radiation therapy is required prior to starting trametinib.
* An interval of at least 48 hours for short-acting colony stimulating factor agents and 10 days interval for long-acting colony stimulating factor agents are required prior to starting trametinib.

  11. Life expectancy Patients must have a life expectancy of greater than 6 months.

  12. Performance level Patients must have a performance status corresponding to a Lansky/Karnofsky score ≥50.

  13. Organ Function Requirements

Participants must have normal organ and marrow function as defined below:

* Total leukocytes ≥ 3,000/µL
* Absolute neutrophil count (ANC) ≥ 1, 000/µL
* Hemoglobin > 80 g/l (transfusion independent within last 2 weeks prior to starting trametinib)
* Platelet count ≥ 100,000/µL (transfusion independent within last 2 weeks prior to starting trametinib)
* Total bilirubin ≤ 1.5 times the ULN within normal institutional limits for age
* Alanine Aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN)*
* Creatinine serum within normal institutional limits for age OR creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
* Creatine phosphokinase ≤ 2x ULN
* A cardiac function defined as Corrected QT (QTcB) interval < 480 msec and LVEF ≥ lower limit of normal (LLN) by echocardiogram (ECHO).
* Blood pressure must be smaller or equal to the 95th percentile for patient's age, height and gender.

  * For uniformity reasons, the ULN for ALT will be 45 U/L in this study

    14. Reproductive status Children of childbearing and child-fathering potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to starting trametinib and for the duration of study participation. Should a female become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Males and females treated or enrolled in this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of trametinib administration. Furthermore, females of childbearing potential (older than 10 years old for this study) must have a negative serum pregnancy test within 7 days prior to starting trametinib. A urine pregnancy test will be done according to evaluation calendar at at 30 days and at 6 months following the last does of study medications.

    15. Administration of oral medication Patients must be able to ingest and retain enterally (per os, nasogastric tube or gastrostomy) administered medication and be free of any clinically significant gastrointestinal abnormalities limiting the absorption of the medication. Tablets cannot be crushed. If the patient cannot swallow tablets, the liquid form should then be used.

SPECIFIC INCLUSION CRITERIA

Participants must belong to one of the following groups to be eligible.

* Group 1: NF1 with Progressing/Refractory LGG (42 patients).
* Group 2: NF1 with Progressing/Refractory PN (46 patients).
* Group 3: Progressing/Refractory LGG with KIAA1549-BRAF fusion (42 patients).
* Group 4: Progressing/Refractory CNS Glioma with activation of the MAPK/ERK pathway who do not meet criteria of other study groups (20 patients).

Exclusion Criteria:

1. Other investigational agents Patients who are receiving any other investigational agents.
2. Cardiac exclusion criteria Patients who have an ejection fraction inferior to the institution LLN, a QTcB ≥ 480 msec or an absolute resting left ventricular ejection fraction (LVEF) of ≤ 39% are not eligible for enrollment.
3. Presence of another malignancy Patient has any other malignancy except if the other primary malignancy is neither currently clinically significant nor requiring active intervention.
4. Previous MEK inhibitor treatment Participants previously treated with a MEK inhibitor who showed less than stable disease during treatment.
5. Tumor with BRAF V600E mutation Patients with a tumor presenting a positive BRAF V600E mutation.
6. Other uncontrollable medical disease Patient has a severe and uncontrollable medical disease (i.e., uncontrolled diabetes, chronic renal disease or active uncontrolled infection), has a chronic liver disease (i.e., chronic active hepatitis and cirrhosis), uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Known HIV infection Patient has a known diagnosis of human immunodeficiency virus (HIV) infection, hepatitis B or C.
8. Previous surgery Patients who had major surgery within 2 weeks prior to starting trametinib.
9. Allergy History of allergic reactions attributed to compounds of similar chemical or biologic composition to trametinib.
10. Previous history of non-compliance Patients with a previous significant history of non-compliance to their treatment or medical regimen.
11. Pregnant or breastfeeding patients Pregnant or breastfeeding female patients are not eligible for this study.

Ages: 1 Month to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 114 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | From date of treatment start until the date of first documented progression, up to completion of treatment (504 treatment days).
  Determination of the objective response rate of daily trametinib as a single agent for treatment of progressing/refractory low-grade tumors with MAPK/ERK pathway activation.

SECONDARY OUTCOMES:
Time to Progression | From date of treatment start up to 3 years following completion of treatment (504 treatment days).
  Time from treatment start, or censored at the date of last disease evaluation for those without progression reported. Applicable to group 1-2-3-4.
Progression Free Survival | From date of treatment start up to 3 years following completion of treatment (504 treatment days).
  Time from treatment start to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at the date of last disease evaluation. Applicable to group 1-2-3-4.
Overall Survival | From date of treatment start up to 3 years following completion of treatment (504 treatment days).
  Time from treatment start to death due to any cause, or censored at date last known alive. Applicable to group 1-2-3-4.
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability). | From treatment start until 30-day follow-up visit.
  Determination of the safety and tolerability of trametinib by assessment of toxicity associated with trametinib (Adverse Events (AEs), Serious Adverse Events (SAEs)). Applicable to group 1-2-3-4.
Determination of the Serum Level of Trametinib. | At Cycle 1 day 22 and at tumor progression OR on Day 1 of Cycle 16 (each cycle is 28 days long).
  Determination of the serum level of trametinib by assessment of the through level. Applicable to group 1-2-3-4.
Evaluation of the Quality of Life During Treatment. | At screening, week 13, week 25, week 37, week 49, week 61 and at the end of treatment day 504.
  Evaluation of the quality of life during treatment with the PedsQL cancer/brain tumor modules. Applicable to group 1-2-3-4.

OTHER OUTCOMES:
Neurocognitive assessment of NF1 patients between 1 and 42 months using the Bayley Scales of Infant and Toddlers Development, Third Edition (Bailey-III). | At study inclusion and at the end of treatment (up to treatment day 504).
  Determine if there are cognitive changes in patients with NF1 during treatment with trametinib. The areas of development assessed to calculate the composite score are: cognition, communication, physical, social/emotional and adaptative. This scale ranges from a score of 40 to 160 with a mean score of 100, where higher scores are desirable.
Neurocognitive assessment of NF1 patients between 2 years and 6 years using the Wechsler Preschool and Primary Scale of Intelligence, Fourth Edition (WPPSI-IV). | At study inclusion and at the end of treatment (up to treatment day 504).
  Determine if there are cognitive changes in patients with NF1 during treatment with trametinib.The areas of cognition assessed to calculate the composite score are: verbal comprehension, visual spatial, fluid reasoning, working memory and processing speed. This scale ranges from a score of 40 to 160 with a mean score of 100, where higher scores are desirable.
Neurocognitive assessment of NF1 patients between 6 years and 16 years and 11 months using the Wechsler Intelligence Scale for Children, Fifth Edition (WISC-V). | At study inclusion and at the end of treatment (up to treatment day 504).
  Determine if there are cognitive changes in patients with NF1 during treatment with trametinib.The areas of cognition assessed to calculate the composite score are: verbal comprehension, visual spatial, fluid reasoning, working memory and processing speed. This scale ranges from a score of 40 to 160 with a mean score of 100, where higher scores are desirable.
Neurocognitive assessment of NF1 patients between 16 years 11 months and 25 years using the Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-IV). | At study inclusion and at the end of treatment (up to treatment day 504).
  Determine if there are cognitive changes in patients with NF1 during treatment with trametinib.The areas of cognition assessed to calculate the composite score are: verbal comprehension, perceptual reasoning, working memory and processing speed. This scale ranges from a score of 40 to 160 with a mean score of 100, where higher scores are desirable.
Response rate of patients with refractory glioma with activation of the MAPK pathway other than BRAF fusion and NF1 | At study inclusion and at the end of treatment (up to treatment day 504).
  Determination of trametinib usefulness in patients with refractory glioma with activation of the MAPK pathway other than BRAF fusion and NF1. Applicable to group 4
Comparison of responses with RECIST 1.1 and volumetric measurement for plexiform neurofibroma | At the achievement of best response to treatment up to treatment day 504.
  Comparison of the best response rate using the RECIST 1.1 criteria and volumetric measurement. Applicable to group 2.
Investigation and correlation of biological features to tumor response. | Within 14 days prior to treatment start for investigations of tumor tissue. At screening, week 13, week 25, week 37, week 49, week 61, at the end of treatment day 504 and every 6 months up to 3 years for ctDNA evaluation.
  Gene expression profiling on fresh frozen tissue and mutational analysis on paraffin-embedded tissue. Circulating tumor DNA (ctDNA) evolution through treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Perreault, MD, Principal Investigator — St. Justine's Hospital
Locations (7):
- Canada (7):
  - Alberta Children's Hospital, Calgary, Alberta
  - Children and Women's Health Centre of British Colombia, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
  - CHU de Québec, Québec, Quebec

REFERENCES:
- [Derived] Perreault S, Larouche V, Tabori U, Hawkin C, Lippe S, Ellezam B, Decarie JC, Theoret Y, Metras ME, Sultan S, Cantin E, Routhier ME, Caru M, Legault G, Bouffet E, Lafay-Cousin L, Hukin J, Erker C, Jabado N. A phase 2 study of trametinib for patients with pediatric glioma or plexiform neurofibroma with refractory tumor and activation of the MAPK/ERK pathway: TRAM-01. BMC Cancer. 2019 Dec 27;19(1):1250. doi: 10.1186/s12885-019-6442-2. PMID 31881853